CLINICAL TRIAL: NCT04282798
Title: Racial Variation in Response to Music Interventions for People With Alzheimer's Dementia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID delay and subsequent unavailability of staff.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00231227
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized Music Intervention (Experimental): Participants will complete a series of questionnaires to identify participants' music preferences and participants' sensitivity to reward from musical engagement. The responses from the music preference questionnaires will be used to create a 1 hr playlist of songs by a member of the study team for the participant to be played daily for four weeks. After playlist is created and transmitted to MP3 device, participants will pick up the equipment and a compliance log will be given for the participant and participants' caregivers to confirm adherence to the protocol of daily listening. The platform will be Spotify, where the MP3 device given to participant at the start of the intervention will be preprogrammed with the participant's personal playlist on the platform. This trial is a supplementary treatment option for cognitive and neuropsychiatric assessments for AD, as such no alterations in the current treatment plans of any participant will be necessary.
  Interventions: Other: Personalized Music Intervention

INTERVENTIONS:
Other: Personalized Music Intervention — Participants will complete a series of questionnaires to identify participants' music preferences and participants' sensitivity to reward from musical engagement. The responses from the music preference questionnaires will be used to create a 1 hr playlist of songs by a member of the study team for the participant to be played daily for four weeks. After playlist is created and transmitted to MP3 device, participants will pick up the equipment and a compliance log will be given for the participant and participants' caregivers to confirm adherence to the protocol of daily listening. The platform will be Spotify, where the MP3 device given to participant at the start of the intervention will be preprogrammed with the participant's personal playlist on the platform. This trial is a supplementary treatment option for cognitive and neuropsychiatric assessments for AD, as such no alterations in the current treatment plans of any participant will be necessary.

SUMMARY:
This project will study the efficacy of a personalized receptive music intervention on neuropsychiatric symptoms and general cognitive function in patients with mild and moderate Alzheimer's disease (AD) by race.

DETAILED DESCRIPTION:
Music interventions have become a popular treatment option to be used alongside medicinal treatment for many chronic conditions including Alzheimer's disease. Healthcare providers and researchers have found that when patients who have chronic conditions engage with music that is patients' preference or most familiar to patients, the patients display positive changes in mood regulation and thinking overall. The investigators are trying to understand to what extent these music interventions could be useful for patients with Alzheimer's disease and for which populations the intervention is more effective for. To do this, the investigators are looking to recruit participants with a diagnosis of Alzheimer's disease to complete a four (4) week personalized music intervention where patients listen to a one-hour playlist created from patients' described preferences and songs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's disease
* English speaking

Exclusion Criteria:

* Deaf or hard of hearing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change in severity of neuropsychiatric symptoms as assessed by the Neuropsychiatric Inventory-Questionnaire (NPI-Q) severity score | Initial and final visit, four weeks apart
  Examining changes in the NPI-Q which is an informant-based interview that assesses 12 neuropsychiatric symptoms of the participant. The NPI-Q includes 12 neuropsychiatric domains. Initial responses to each domain question are "Yes" (present) or "No" (absent). If the response to the domain question is "No", the informant goes to the next question. If "Yes", the informant then rates the severity of the symptoms present on a 3-point scale where 1 is "mild" and 3 is "severe".
Change in Montreal Cognitive Assessment (MoCA) score | Initial and final visit, four weeks apart
  Examining changes in the MoCA which is a cognitive test for Alzheimer's disease. The MoCA assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation to time and place. MoCA total scores range between 0 and 30; 18-25 = mild cognitive impairment, 10-17 = moderate cognitive impairment and less than 10 = severe cognitive impairment.

SECONDARY OUTCOMES:
Correlation between the Barcelona Music Reward Questionnaire (BMRQ) score and NPI-Q score | At the end of the study, up to 9 months
  The 20-item Barcelona Music Reward Questionnaire (administered at enrollment) assesses facets of the music and reward experiences with 5 factors: Musical Seeking, Emotion Evocation, Mood Regulation, Social Reward, and Sensory-Motor. Participants indicate the level of agreement with each statement by using a five-point scale ranging from ''fully disagree'' (1) to ''fully agree'' (5). BMRQ total scores range between 20 and 100. BMRQ total scores and NPI-Q totals scores will be used to assess whether these variables correlate. The correlation will be completed via statistical analysis in a chi squared test.
Correlation between the BMRQ score and MoCA score | At the end of the study, up to 9 months
  The 20-item BMRQ (administered at enrollment) assesses facets of the music and reward experiences with 5 factors: Musical Seeking, Emotion Evocation, Mood Regulation, Social Reward, and Sensory-Motor. Participants indicate the level of agreement with each statement by using a five-point scale ranging from ''fully disagree'' (1) to ''fully agree'' (5). BMRQ total scores range between 20 and 100. BMRQ total scores and MoCA total scores will be used to assess whether these variables correlate. The correlation will be completed via statistical analysis in a chi squared test.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Rosenberg, MD, Principal Investigator — Johns Hopkins University; Melissa K Eustache, BS, Study Director — Johns Hopkins University Kreiger School of Arts & Sciences